CLINICAL TRIAL: NCT04993768
Title: A Phase 2a Study of TPN-101 in Patients With Progressive Supranuclear Palsy (PSP)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Transposon Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TPN-101-PSP-201
Record Dates: First submitted 2021-07-19; First posted 2021-08-06 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Progressive Supranuclear Palsy
MeSH Terms: conditions — Supranuclear Palsy, Progressive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TPN-101, Dose A (Experimental)
  Interventions: Drug: TPN-101, 100 mg/day
- TPN-101, Dose B (Experimental)
  Interventions: Drug: TPN-101, 200 mg/day
- TPN-101, Dose C (Experimental)
  Interventions: Drug: TPN-101, 400 mg/day
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TPN-101, 100 mg/day — 100 mg/day of study investigational drug TPN-101 once daily for 24 weeks (double-blind treatment) followed by 400 mg/day TPN-101 for 24 weeks (open-label treatment).
  Arms: TPN-101, Dose A
Drug: TPN-101, 200 mg/day — 200 mg/day of study investigational drug TPN-101 once daily for 24 weeks (double-blind treatment) followed by 400 mg/day TPN-101 for 24 weeks (open-label treatment).
  Arms: TPN-101, Dose B
Drug: TPN-101, 400 mg/day — 400 mg/day of study investigational drug TPN-101 once daily for 24 weeks (double-blind treatment) followed by 400 mg/day TPN-101 for 24 weeks (open-label treatment).
  Arms: TPN-101, Dose C
Drug: Placebo — Placebo once daily for 24 weeks (double-blind treatment) followed by 400 mg/day TPN-101 for 24 weeks (open-label treatment).
  Arms: Placebo

SUMMARY:
This is a Phase 2a study to assess the safety and tolerability of TPN-101 patients with PSP.

DETAILED DESCRIPTION:
This is a Phase 2a multi-center, randomized, double-blind, placebo-controlled parallel-group, 4-arm study with an open-label treatment phase in patients with PSP. This study includes a 6-week Screening Period, a 24-week Double-blind Treatment Period, a 24-week Open label Treatment Period, and a Follow-up Visit 4 weeks post treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of probable progressive supranuclear palsy (PSP)
2. Presence of PSP symptoms for less than 5 years
3. Has a reliable caregiver/informant to accompany the patient to all study visits.
4. Score ≥ 18 on the Mini Mental State Exam (MMSE) at Screening
5. Patient must reside outside a skilled nursing facility or dementia care facility at the time of Screening, and admission to such a facility must not be planned. Residence in an assisted living facility is allowed

Exclusion Criteria:

Patients must not meet any of the following criteria:

1. Presence of other significant neurological or psychiatric disorders
2. History of clinically significant brain abnormality
3. Presence of cerebellar ataxia, choreoathetosis, early symptomatic autonomic dysfunction, or moderate to severe resting tremor, responsive to levodopa
4. Known history of serum or plasma progranulin level less than one standard deviation below the normal patient mean
5. Known presence of disease-associated mutation in TARDBP, GRN, CHMPB2, or VCP genes; or any other frontotemporal lobar degeneration causative genes not associated with underlying tau pathology
6. History of clinically significant hematological, endocrine, cardiovascular, renal, hepatic, or gastrointestinal disease

Ages: 41 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess the safety and tolerability of TPN-101 in patients with progressive supranuclear palsy (PSP) | 48 weeks
  Incidence and severity of spontaneously reported treatment-emergent adverse events (TEAEs) associated with TPN-101 v. placebo administered for up to 48 weeks in patients with PSP

SECONDARY OUTCOMES:
Assess the pharmacokinetics of TPN-101 as measured by concentrations of TPN-101 in plasma and cerebrospinal fluid (CSF) | 48 weeks
Assess the pharmacodynamic effect of TPN-101 on neurodegeneration as measured by changes in the levels of CSF and blood neurofilament light (NfL) | 48 weeks
Assess the clinical effect of TPN-101 as measured by changes in score on the Progressive Supranuclear Palsy Rating Scale (PSPRS) | 48 weeks
  The PSPRS is comprised of 28 items in six categories: daily activities (by history), behavior, bulbar, ocular motor, limb motor and gait/midline. Scores range from 0 to 100, each item is graded 0-2 (six items) or 0-4 (22 items), with lower scores indicating better clinical and functional status.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - St. Joseph's Hospital and Medical Center, Barrow Neurological Institute, Phoenix, Arizona
  - UC San Diego Altman Clinical And Translational Research Institute, La Jolla, California
  - UCSF Neurosciences Clinical Research Unit (NCRU), San Francisco, California
  - Rocky Mountain Movement Disorders Center, Englewood, Colorado
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - UFHealth Fixel Institute for Neurological Diseases, Gainesville, Florida
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Irving Center for Clinical and Translational Research, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas